CLINICAL TRIAL: NCT01660217
Title: Eczema Action Plan Improves Patient and Caregiver Understanding and Perception of Atopic Dermatitis Management: A Randomized Controlled Trial
Brief Title: Eczema Action Plan Improves Patient and Caregiver Understanding and Perception of Atopic Dermatitis Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dermatology & Aesthetics of Wicker Park (Other)
Responsible Party: Principal Investigator, Peter A. Lio, MD, Attending Physician in Dermatology, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: EAP-1
Record Dates: First submitted 2012-07-31; First posted 2012-08-08 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; eczema action plan; patient education; written handout; investigator's global assessment; randomized controlled trial
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Initial Verbal Instruction Group (Experimental): The group who initially received only verbal instruction, and then later (in the "crossover portion") received a written Eczema Action Plan (EAP)
  Interventions: Other: A written Eczema Action Plan (EAP)
- Written Eczema Action Plan (EAP) (Experimental): The group given a written EAP after verbal instruction
  Interventions: Other: A written Eczema Action Plan (EAP)

INTERVENTIONS:
Other: A written Eczema Action Plan (EAP) — A written Eczema Action Plan (EAP) was given to the patients with their treatment regimen.

SUMMARY:
This is a randomized controlled study. The control group will consist of adult subjects and the caregivers of pediatric subjects with an established diagnosis of atopic dermatitis (AD), who are visiting a dermatologist for a standard AD office visit. In the control group, only verbal instruction (VI), the standard of care, will be provided. The intervention group will receive a similar VI with an additional component: an eczema education handout, as well as an individualized written Eczema Action Plan (EAP) that will illustrate how to recognize disease flare-ups and subsequent remissions. In addition, the EAP will provide detailed step-wise instructions regarding treatment modifications for the above-mentioned variations in treatment severity. To ensure that all patients ultimately receive the same level of care, the control group will also receive an EAP at the end of their consultation.

The goal of this study is to assess subjects' perception in the provider's use of an EAP and its effectiveness in helping patients understand their disease and management plan. In order to evaluate the primary end-points, subjects in both the control and treatment groups will be asked to complete post-consultation surveys. Four post-consultation outcomes will be measured: (1) caregivers' understanding of the disease and treatment, (2) caregivers' comfort level in following the EAP at home, (3) caregivers' anxiety level in managing the AD at home, and (4) caregivers' preference for VI + EAP as compared to VI alone, EAP alone, or neither the EAP nor the VI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older fulfilling Hanifin and Rajka diagnostic criteria for AD, or adult caregivers for patients younger than 18 years of age, and the ability to comprehend study materials in English

Exclusion Criteria:

* Prior exposure to written action plans

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Participants understanding of atopic dermatitis and homecare regimen | At the beginning of the visit and at the end of the visit (approximately 45min later)

SECONDARY OUTCOMES:
Changes in emotional distress level on disease self-management | At the beginning of the visit and at the end of the visit (approximately 45min later)

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology & Aesthetics of Wicker Park, Chicago, Illinois, United States